CLINICAL TRIAL: NCT04623463
Title: Effects of Physical Activity on OSA Severity Based on the Level of Fluid Shift in Patients Who Can't Use CPAP or MAD
Brief Title: Effects of Physical Activity on OSA Severity Based on the Level of Fluid Shift
Acronym: AP-FLUID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: HP2 Laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC20.105
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise intervention (Other): Participants included in the present study will benefit from a 4-week physical activity intervention. Upon the initial visit, a physical activity prescription will be defined and they will be equipped with a physical activity monitor that allows feedback. Participants will then exercise one day per week on-site and 4 days/week on their own. Weekly physical activity will be reviewed weekly with the participant during their on-site visit.
  Interventions: Behavioral: Physical activity intervention

INTERVENTIONS:
Behavioral: Physical activity intervention — Participants included in the present study will benefit from a 4-week physical activity intervention. Upon the initial visit, a physical activity prescription will be defined and they will be equipped with a physical activity monitor that allows feedback. Participants will then exercise one day per week on-site and 4 days/week on their own. Weekly physical activity will be reviewed weekly with the participant during their on-site visit.

SUMMARY:
Obstructive sleep apnea (OSA) is characterized by complete or partial upper-airway collapse during sleep associated with sleepiness. OSA causes severe impairments in quality of life (sleepiness, tiredness, concentration difficulties). Moreover, OSA has adverse consequences on the cardiovascular system by causing intermittent hypoxia, increased sympathetic nervous system activation and vascular endothelial dysfunction.

Continuous Positive Airway Pressure (CPAP) and mandibular advanced devices (MAD) remain the two first-line therapies for OSA. However, not all patients are eligible for these treatments or are not able to follow for a lifelong therapy and therefore do not use it consistently.

A recent meta-analysis has confirmed that regular physical activity reduces OSA by approximately 28% (Mendelson et al. 2018). However, an important inter-individual variability exists and no study to date has identified characteristics of patients who respond to these interventions.

The aim of this Prospective study, single-site, non-randomized 4-week trial is to evaluate the impact of a 4-week physical activity intervention on the apnea-hypopnea index (AHI) in OSA patients based on their baseline fluid shift level.

Participants included in the present study will benefit from a 4-week physical activity intervention. Upon the initial visit, a physical activity prescription will be defined and they will be equipped with a physical activity monitor that allows feedback. Participants will then exercise one day per week on-site and 4 days/week on their own. Weekly physical activity will be reviewed weekly with the participant during their on-site visit.

ELIGIBILITY:
Inclusion Criteria:

* • Patient aged 18 to 80 years old

  * Patient with OSA (AHI ≥ 15 events/hr)
  * Patient not receiving any treatment for their OSA
  * Patient able to provide written informed consent
  * Patient able to participate in regular physical activity (no medical contraindication to exercise)

Exclusion Criteria:

* • Pregnancy

  * Person deprived of liberty or subject to a legal protection measure
  * Patient presenting a condition that can influence the results. (According to the investigator's judgment, i.e. heart failure, venous insufficiency).
  * Vulnerable person or legally protected adult.
  * Patients already included in another interventional study
  * BMI > 30 kg/m²
  * Patient taking diuretics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea index | Baseline-4weeks
  Measured during polysomnography

SECONDARY OUTCOMES:
Subjective sleepiness as measured by the Epworth Sleepiness Score | Baseline-4weeks
  Measured with the Epworth Sleepiness Score Questionnaire
Overnight change in leg fluid volume | Baseline-4weeks
  Measured using bio-electrical impedance
Quality of life assessed by the SF-36 questionnaire | Baseline-4weeks
  Measured using the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- UniversityGrenobleHospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided